CLINICAL TRIAL: NCT04631094
Title: Nurse, PhD Student, Responsible Researcher
Brief Title: The Effect of Two Different Structured Balls on Pain and Fear Levels During Venous Blood Collection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Yurdakul (Other)
Responsible Party: Sponsor-Investigator, Zeynep Yurdakul, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pediatric Nursing
Record Dates: First submitted 2020-10-24; First posted 2020-11-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Nurse's Role
Keywords: child, fear, nursing, pain, venipuncture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The results were planned by the statistician as the evaluator and the experts who will score the video recording, blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): The group holding the serrated ball in the hand on the extremity from which venous blood will be taken
  Interventions: Other: The group holding the serrated ball in the hand on the extremity from which venous blood will be taken
- Group 2 (Experimental): The group holding the serrated ball in the hand on the opposite side of the extremity from which venous blood will be taken.
  Interventions: Other: The group holding the serrated ball in the hand on the opposite side of the extremity from which venous blood will be taken.
- Group 3 (Experimental): The group holding a smooth ball in the hand on the extremity from which venous blood will be taken
  Interventions: Other: The group holding a smooth ball in the hand on the extremity from which venous blood will be taken
- Group 4 (Experimental): The group holding a smooth ball in the hand opposite the extremity from which venous blood will be taken.
  Interventions: Other: The group holding a smooth ball in the hand opposite the extremity from which venous blood will be taken.
- Group 5 (No Intervention): The group that will undergo standard hospital blood collection procedure.

INTERVENTIONS:
Other: The group holding the serrated ball in the hand on the extremity from which venous blood will be taken — Children in the experimental groups will squeeze the serrated ball during the blood draw.
  Other Names: serrated ball
  Arms: Group 1
Other: The group holding the serrated ball in the hand on the opposite side of the extremity from which venous blood will be taken. — Children in the experimental groups will squeeze the serrated ball during the blood draw.
  Other Names: serrated ball
  Arms: Group 2
Other: The group holding a smooth ball in the hand on the extremity from which venous blood will be taken — Children in the experimental groups will squeeze the smooth ball during the blood draw.
  Other Names: smooth ball
  Arms: Group 3
Other: The group holding a smooth ball in the hand opposite the extremity from which venous blood will be taken. — Children in the experimental groups will squeeze the smooth ball during the blood draw.
  Other Names: smooth ball
  Arms: Group 4

SUMMARY:
Pain causes many physiological and psychological changes in the body, increases the level of anxiety in children, and prolongs examination and other procedures. Pain should be evaluated individually for each child, taking into account individual differences in pain level and response to pain. From the moment of birth, human beings have been exposed to many invasive interventions throughout their lives and experience pain and anxiety as a result. Experiences with childhood pain shape children's future pain responses.

This study, which was planned to stimulate the touch receptors of two different balls used during venous blood collection, is a randomized controlled study in order to determine the effect on the pain and fear levels of children aged 6-12 years. A total of 310 children were included in the study. The experimental groups included in the study were asked to hold the balls with their hands according to their groups, no attempt was made to the control group. The research data were obtained with the Wong-Baker Faces Pain Rating Scale and Child Fear Scale, which will be used in the evaluation. In addition, oxygen saturation and heart rate were evaluated immediately before and after removal of the tourniquet.

DETAILED DESCRIPTION:
Attempt During the trial, all blood collection procedures will be performed by the same nurse working in the hospital's blood collection unit. The nurse who will perform the procedure works as a pediatric nurse for 15 years.

Control Group;

* Data on the child and his parents will be collected by the researcher using face-to-face interview technique and recorded in the "Information Form".
* The child and parent will be informed by showing the Wong-Baker Faces Pain Rating Scale, the Child Fear Scale, and the pulse oximeter.
* Disinfectant will be poured on the child's and parent's hands.
* Before the blood draw, the child will be given the Wong-Baker Faces Pain Rating Scale, the Child Fear Scale, and a pen, and will be asked to mark the facial expression appropriate to his current situation.
* The child who filled out the form will be taken to the blood collection room with his parents, and the child will be seated on the blood collection chair. The child and parent will be informed about the blood collection procedure according to the hospital procedure.
* Due to the pandemic, in accordance with the hospital procedure, the tourniquet will be disinfected and used after each blood collection.
* The nurse will determine the child's extremity suitable for vascular access.
* Standard hospital procedures will be applied throughout the blood collection procedure.
* Immediately after the procedure, the child will be asked to mark the appropriate facial expression on the Wong-Baker Faces Pain Rating Scale and the Child Fear Scale during the procedure.
* Disinfectant will be poured on the child's and parent's hands.
* The child whose blood collection process is completed, and his parents will be thanked for their acceptance to participate in the research and will be ensured to leave the room.

Experimental Groups;

* Data on the child and his parents will be collected by the researcher using face-to-face interview technique. It will be saved in the "Information Form".
* The child and parent will be informed by showing the Wong-Baker Faces Pain Rating Scale, the Child Fear Scale, and the pulse oximeter.
* Disinfectant will be poured on the child's and parent's hands.
* Before the blood draw, the child will be given the Wong-Baker Faces Pain Rating Scale, the Child Fear Scale, and a pen, and will be asked to mark the facial expression appropriate to his current situation.
* The child who filled out the form will be taken to the blood collection room with his parents, and the child will be seated on the blood collection chair. The child and parent will be informed about the blood collection procedure according to the hospital procedure.
* Due to the pandemic, in accordance with the hospital procedure, the tourniquet will be disinfected and used after each blood collection.
* The nurse will determine the child's extremity suitable for vascular access.
* According to randomization, the child was able to hold the ball according to the group (Group 1, Group 2, Group 3, Group 4).

  * Group 1: Serrated ball + extremity group from which venous blood will be taken
  * Group 2: Serrated ball + hand group on the opposite side of the extremity from which venous blood will be taken
  * Group 3: Straight ball + extremity group from which venous blood will be taken
  * Group 4: Flat ball + hand group on the opposite side of the extremity from which venous blood will be taken
  * Control group: Group to be applied standard hospital blood collection procedure
* Standard hospital procedures will be applied throughout the blood collection procedure.
* Immediately after the procedure, the child will be asked to mark the appropriate facial expression on the Wong-Baker Faces Pain Rating Scale and the Child Fear Scale during the procedure.
* Disinfectant will be poured on the child's and parent's hands.
* The child whose blood collection process is completed, and his parents will be thanked for their acceptance to participate in the research and will be ensured to leave the room.

ELIGIBILITY:
Inclusion Criteria:

* - The volunteerism of the child and the parent to participate in the research,
* The child is between the ages of 5-12,
* The child and the parent speaks Turkish, Taking blood from the cephalic vein,
* Turnstile not being tied for more than 30 seconds,
* Not taking any analgesic (systemic or topical), antipyretic, anti-inflammatory drugs in the last 12 hours,
* Body temperature between 36.5-37.2 ⁰C,
* Not having a disease that can cause chronic pain,
* No acute pain or anxiety during the procedure,
* Absence of skin integrity problems,
* No obstacle to grip the balls in hand,
* Children who do not have regular invasive interventions (no chronic diseases that require blood control such as cancer, diabetes),
* Blood collection was performed at the first attempt,
* The child does not have any auditory, mental or neurological disability that will affect his participation in the research.

Exclusion Criteria:

* - The child and the parents are not willing to participate in the research,
* The child is not between the ages of 5-12,
* The child and the parent do not speak Turkish, Inability to take blood from the cephalic vein,
* Turnstile remaining tied for more than 30 seconds,
* Taking any medication with analgesic (systemic or topical), antipyretic or anti-inflammatory effects in the last 12 hours,
* Body temperature lower than 36.5 C-37.2 ⁰C,
* Having a disease that can cause chronic pain,
* Children who undergo regular invasive interventions (having chronic diseases that require blood control such as cancer, diabetes), Failure to take blood at the first attempt,
* Any acute pain or anxiety during the procedure,
* Problems with skin integrity,
* It has an obstacle to grip the balls,
* Having an auditory, mental or neurological disability that will affect the child's participation in the research,
* Children in the control group want or involuntarily hold their parent's hand or something else during the procedure.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 310 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain level as assessed with Wong-Baker Faces Pain Rating Scale | during the procedure
  This scale to be used to assess pain in our study was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983. The scale is widely used to measure pain intensity in children over the age of three. Pain is scored according to numerical values assigned to faces that show an expression spectrum; smiling face represents no pain (0 points), crying face represents severe pain (10 points). The scale is a valid and reliable tool for measuring procedural pain severity. Permission for the scale was obtained from the official website of the Wong-Baker Faces Foundation. The Turkish translation of the scale was sent by Nick Baker, official site official of the Wong-Baker Faces Foundation.
Fear as assessed using the Child Fear Scale | during the procedure
  It is used to determine the child's fear and anxiety level. Fear and anxiety are assessed on a five-point scale. The single-item scale consists of five facial expressions regardless of gender. The first facial expression of the scale is neutral and has a value of zero. The last facial expression is worth four points expressing extreme fear. In this study, Child Fear Scale will be used to evaluate the fear levels of children in the experimental and control groups before and after the bloodletting procedure. The scale was introduced into the Turkish language by Gerçeker et al. (2018). Test-retest reliability of the Child Fear Scale was found to be quite high, and its content validity index was determined as 0.89. Since the scale is in the form of scoring, item-total correlation and Cronbach alpha coefficient could not be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Işık ESENAY, Study Director — assistant professor
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The child is between the ages of 6-12,
  * Volunteering of the child and parent to participate in the research,
  * Acceptance of wearing the transparent mask provided by the researcher, which clearly shows the facial expression, throughout the procedure,
  * Turkish speaking of the child and the parent,
  * The child does not have an auditory, mental or neurological disability that will affect his participation in the research,
  * Absence of problems related to skin integrity on the hand,
  * There is no obstacle to the grasp of the balls,
  * Not taking analgesic (systemic or topical), antipyretic, anti-inflammatory drugs in the last 12 hours,
  * Body temperature between 36.5-37.2 ⁰C,
  * Absence of acute pain before the procedure,
  * Absence of a disease that may cause chronic pain,
  * No regular invasive intervention (no chronic disease requiring blood control such as cancer, diabetes).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: always
Access Criteria: Considering that repeated attempts may increase pain and anxiety in children, blood sampling cannot be performed in the first attempt,
  * Children in the control group wanting or involuntarily holding their parents' hand or anything during the procedure,
  * Failure to enter the vein within 20 seconds of grasping the ball,
  * Failure to take blood from the cephalic vein,
  * The children in the experimental group let go of the ball in their hands during the procedure.